CLINICAL TRIAL: NCT05339750
Title: Democratization of Allergy Skin Patch Testing to Increase Efficiency and Scale of the Practice
Brief Title: Allergy Skin Patch Artificial Intelligence (AI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Matthew Hall, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 21-011596
Record Dates: First submitted 2022-04-04; First posted 2022-04-21 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Allergic Contact Dermatitis
MeSH Terms: conditions — Dermatitis, Allergic Contact

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Allergy Skin Patch Testing (Experimental): On day 1, subjects will have a allergy skin patch test applied and a routine skin examination. On day 3, the patch test will be removed and documentation of the test sites using iPhone app. On day 5, the final assessment for allergic contact dermatitis will be conducted by a medical professional.
  Interventions: Device: AI-based smartphone application; Diagnostic Test: Allergen patch

INTERVENTIONS:
Device: AI-based smartphone application — AI-based smartphone application to record and interpret the patch test results
Diagnostic Test: Allergen patch — Allergens applied to a patch which is placed on the skin on the forearm region. The patch contains 10 dime-sized disks which contain a different allergen.

SUMMARY:
The purpose of this research is to assess human and artificial intelligence performance in grading contact dermatitis reactions in healthy volunteers.

DETAILED DESCRIPTION:
Study participation involves three visits to the study site on Days 1, 3, and 5, and completion of a demographics and allergy history questionnaire. Researchers will review medical history and current medications. On Day 1 a patch will be applied with 10 allergens and a routine skin examination will be conducted and a photograph will be taken of the forearm. On day 3, subjects will return to remove the patch test and have photographs of the area taken. On day 5, the final assessment for allergic contact dermatitis will be performed and photographs of the area taken.

Key Information: The most common side effect of skin testing is slightly swollen, red, itchy bumps (wheals). These wheals may be most noticeable during the test. In some, an area of swelling, redness and itching may develop a few hours after the test and remain for a couple of days. Rarely, allergy skin tests can produce a severe, immediate allergic reaction. The patches are worn on the forearm for 48 hours. During this time, bathing and activities that cause heavy sweating should be avoided. Irritated skin at the patch site may indicate an allergy. If a positive test result is documented, a medical professional will provide education and recommend follow up with primary care provider.

ELIGIBILITY:
Inclusion Criteria

* Adults over the age of 18
* Willing and able to provide informed consent

Exclusion Criteria

* Under 18 years of age
* Has used topical or oral steroids two weeks prior to patch testing
* Currently taking immunosuppression agents or is immunocompromised due to medical condition
* No sunburn or rash at site of testing
* Women who are breastfeeding or pregnant.
* Treatment with ultraviolet (UV) light (including tanning) during the two weeks prior to visit.
* Subjects unable to comply with patch test study requirements including multiple return visits and activity restrictions (e.g., protecting patch test area from excess moisture due to showering)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2022-09-23 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
AI algorithms predictions of reactions | 6 months
  Number of times the AI algorithms matches the human review of photographs of skin patch tests classification of reaction. The accuracy for the classification of regions within the test panel that either were a reaction (reaction grade 1+) or not (grade 0).

SECONDARY OUTCOMES:
Fitzpatrick skin type assessment | 10 months
  Number of times the AI algorithms matches the human review of photographs of skin patch tests over the entire range of Fitzpatrick skin types. The Fitzpatrick skin typing categorize skin type according to how much melanin is present.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Hall, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials